CLINICAL TRIAL: NCT06813170
Title: Diet With or Without Metarecod® in Obese Subjects With Type 2 Diabetes: Effect on Body Weight, in Vivo Oxidative Stress, Endothelial Function, Low-grade Inflammation and Gut Microbiota
Brief Title: Diet With or Without Metarecod® in Obese Subjects With Type 2 Diabetes
Acronym: MONDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6264
Record Dates: First submitted 2025-01-15; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metarecod + Diet (Experimental): Patients will be given diet and they will take Metarecod 1 sachet twice daily. The diet program will be calculated to achieve a 20% caloric relative decrease from habitual intake, for an average energy deficit of 500 kcal/daily
  Interventions: Dietary Supplement: Metarecod; Other: Diet
- Low caloric diet (Placebo Comparator): Patients will be given diet program calculated to achieve a 20% caloric relative decrease from habitual intake, for an average energy deficit of 500 kcal/daily with <30% of total calories from fat and at least 15% from proteins.
  Interventions: Other: Diet

INTERVENTIONS:
Dietary Supplement: Metarecod — Policaptil Gel Retard: Metarecod®. The medical device will be given as 1 sachet twice daily
  Arms: Metarecod + Diet
Other: Diet — Diet program will be planned to achieve a ≥8% body weight relative reduction over 12 months and tailored calculating a 20% caloric relative decrease from habitual energy intake, corresponding to an average energy deficit of approximately 500 kcal/daily (approximately a total of 1,200-1,500/daily Kcal for women and 1,500-1,800/daily Kcal for men), with <30% of total calories from fat (<10% from satured fats) and at least 15% of total calories from proteins. For carbohydrate intake, low glycemic index food will be preferred to high glycemic index food, to prevent higher post prandial glycemic excursions

SUMMARY:
Obesity is considered the largest chronic non-communicable disease (globesity) worldwide with a growing trend in the near future. Weight loss programs are strongly recommended in obese patients, especially with type 1 diabetes mellitus (T2DM), although the majority of subjects do not reach or maintain the recommended weight loss target with nutritional intervention alone and one-third of those who achieve a significant weight loss returns to original body weight within one year. Metarecod® (Neopolicaptil Gel Retard) is a substance based medical device consisting of a macromolecule complex derived from high-fiber raw materials, whose mode of action consists in creating an endoluminal gel in the gut that limits glucose and lipids absorption. The primary aim of the present study is to assess whether the combination of Metarecod® and standard diet as compared to diet alone can achieve a superior weight loss over 12 months of treatment. The present study will also compare the effects of the combination of Metarecod® and diet vs diet alone on:

1. the improvement of glycemic variability and metabolic indexes;
2. the oxidative status, the endothelial anti-thrombotic activity, the inflammatory status;
3. the induction of favorable changes in gut microbiota composition and intestinal permeability.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent at study entry;
2. Age: 30-70 years;
3. T2DM diagnosis according to the American Diabetes Association criteria since ≥6 months;
4. Stable metabolic control as indicated by levels of glycated hemoglobin (HbA1c) <7.5% on two consecutive measurements before study enrollment;
5. Body mass index (BMI) level ≥30 Kg/m2 during the 3 months preceding randomization.

Exclusion Criteria:

1. Chronic treatment with corticosteroids and/or chronic treatment with non-steroidal inflammatory drugs, defined as ≥3 times/week with the rationale that these drugs independently impact on the whole inflammatory state;
2. Clear indication for dual antiplatelet therapy and/or anticoagulant therapy (full dose);
3. Active cancer or cancer in complete remission from less than one year, except for treated early-stage squamous or basal cell skin carcinomas;
4. For women with childbearing potential, pregnancy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 12 months
  Difference in body weight expressed in kg after 12 months between randomized arms

SECONDARY OUTCOMES:
Glycemic variability | 12 months
  Glycemic variability, as assessed by continuous glucose monitoring (CGM)
8-iso-Prostaglandin (PG) F2α | 12 months
  Change on the oxidative status in vivo, as assessed by the measurement of the urinary excretion of the F2-isoprostane
2,3-dinor-6-keto-PGF1α | 12 months
  Change of the endothelial anti-thrombotic activity in vivo as assessed by the production of the vasodilator and platelet inhibitor prostanoid, prostacyclin (PGI2), major urinary enzymatic metabolite 2,3-dinor-6-keto-PGF1α
Interleukin (IL)-6 | 12 months
  Change on inflammatory status assessed through the change of serum levels of interleukin (IL-6)
C-reactive protein | 12 months
  Change on inflammatory status assessed through the change of serum levels of C-reactive protein (CRP)
Waist circumference | 12 months
  Change in waist circumference after 12 months between arms
Achieving the target weight loss | 12 months
  Percentage of subjects who will reach the target percentage weight loss of 8%
Gut microbiota composition | 12 months
  Gut microbiota composition, assessed by 16S RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Dario Pitocco, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS; UOC Diabetologia, Rome, Lazio, Italy

REFERENCES:
- [Background] Danne T, Nimri R, Battelino T, Bergenstal RM, Close KL, DeVries JH, Garg S, Heinemann L, Hirsch I, Amiel SA, Beck R, Bosi E, Buckingham B, Cobelli C, Dassau E, Doyle FJ 3rd, Heller S, Hovorka R, Jia W, Jones T, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Maahs D, Murphy HR, Norgaard K, Parkin CG, Renard E, Saboo B, Scharf M, Tamborlane WV, Weinzimer SA, Phillip M. International Consensus on Use of Continuous Glucose Monitoring. Diabetes Care. 2017 Dec;40(12):1631-1640. doi: 10.2337/dc17-1600. PMID 29162583
- [Background] Rocca B, Tosetto A, Betti S, Soldati D, Petrucci G, Rossi E, Timillero A, Cavalca V, Porro B, Iurlo A, Cattaneo D, Bucelli C, Dragani A, Di Ianni M, Ranalli P, Palandri F, Vianelli N, Beggiato E, Lanzarone G, Ruggeri M, Carli G, Elli EM, Carpenedo M, Randi ML, Bertozzi I, Paoli C, Specchia G, Ricco A, Vannucchi AM, Rodeghiero F, Patrono C, De Stefano V. A randomized double-blind trial of 3 aspirin regimens to optimize antiplatelet therapy in essential thrombocythemia. Blood. 2020 Jul 9;136(2):171-182. doi: 10.1182/blood.2019004596. PMID 32266380
- [Background] Zaccardi F, Rizzi A, Petrucci G, Ciaffardini F, Tanese L, Pagliaccia F, Cavalca V, Ciminello A, Habib A, Squellerio I, Rizzo P, Tremoli E, Rocca B, Pitocco D, Patrono C. In Vivo Platelet Activation and Aspirin Responsiveness in Type 1 Diabetes. Diabetes. 2016 Feb;65(2):503-9. doi: 10.2337/db15-0936. Epub 2015 Oct 15. PMID 26470782
- [Background] Santilli F, Zaccardi F, Liani R, Petrucci G, Simeone P, Pitocco D, Tripaldi R, Rizzi A, Formoso G, Pontecorvi A, Angelucci E, Pagliaccia F, Golato M, De Leva F, Vitacolonna E, Rocca B, Consoli A, Patrono C. In vivo thromboxane-dependent platelet activation is persistently enhanced in subjects with impaired glucose tolerance. Diabetes Metab Res Rev. 2020 Feb;36(2):e3232. doi: 10.1002/dmrr.3232. Epub 2019 Nov 15. PMID 31671234
- [Background] Tanase DM, Gosav EM, Neculae E, Costea CF, Ciocoiu M, Hurjui LL, Tarniceriu CC, Maranduca MA, Lacatusu CM, Floria M, Serban IL. Role of Gut Microbiota on Onset and Progression of Microvascular Complications of Type 2 Diabetes (T2DM). Nutrients. 2020 Dec 2;12(12):3719. doi: 10.3390/nu12123719. PMID 33276482
- [Background] Badimon L, Vilahur G, Rocca B, Patrono C. The key contribution of platelet and vascular arachidonic acid metabolism to the pathophysiology of atherothrombosis. Cardiovasc Res. 2021 Jul 27;117(9):2001-2015. doi: 10.1093/cvr/cvab003. PMID 33484117
- [Background] Roest M, Voorbij HA, Van der Schouw YT, Peeters PH, Teerlink T, Scheffer PG. High levels of urinary F2-isoprostanes predict cardiovascular mortality in postmenopausal women. J Clin Lipidol. 2008 Aug;2(4):298-303. doi: 10.1016/j.jacl.2008.06.004. Epub 2008 Jun 13. PMID 21291746
- [Background] Petrucci G, Zaccardi F, Giaretta A, Cavalca V, Capristo E, Cardillo C, Pitocco D, Porro B, Schinzari F, Toffolo G, Tremoli E, Rocca B. Obesity is associated with impaired responsiveness to once-daily low-dose aspirin and in vivo platelet activation. J Thromb Haemost. 2019 Jun;17(6):885-895. doi: 10.1111/jth.14445. Epub 2019 Apr 29. PMID 30933424
- [Background] Patrono C, FitzGerald GA. Isoprostanes: potential markers of oxidant stress in atherothrombotic disease. Arterioscler Thromb Vasc Biol. 1997 Nov;17(11):2309-15. doi: 10.1161/01.atv.17.11.2309. PMID 9409197
- [Background] Guarino G, Della Corte T, Strollo F, Gentile S; Nefrocenter Research Study Group. Policaptil Gel Retard in adult subjects with the metabolic syndrome: Efficacy, safety, and tolerability compared to metformin. Diabetes Metab Syndr. 2021 May-Jun;15(3):901-907. doi: 10.1016/j.dsx.2021.03.032. Epub 2021 Apr 8. PMID 33906073
- [Background] Stagi S, Lapi E, Seminara S, Pelosi P, Del Greco P, Capirchio L, Strano M, Giglio S, Chiarelli F, de Martino M. Policaptil Gel Retard significantly reduces body mass index and hyperinsulinism and may decrease the risk of type 2 diabetes mellitus (T2DM) in obese children and adolescents with family history of obesity and T2DM. Ital J Pediatr. 2015 Feb 15;41:10. doi: 10.1186/s13052-015-0109-7. PMID 25774705
- [Background] Fornari E, Morandi A, Piona C, Tommasi M, Corradi M, Maffeis C. Policaptil Gel Retard Intake Reduces Postprandial Triglycerides, Ghrelin and Appetite in Obese Children: A Clinical Trial. Nutrients. 2020 Jan 14;12(1):214. doi: 10.3390/nu12010214. PMID 31947628
- [Background] Petrucci G, Rizzi A, Hatem D, Tosti G, Rocca B, Pitocco D. Role of Oxidative Stress in the Pathogenesis of Atherothrombotic Diseases. Antioxidants (Basel). 2022 Jul 20;11(7):1408. doi: 10.3390/antiox11071408. PMID 35883899
- [Background] Canuto R, Garcez A, de Souza RV, Kac G, Olinto MTA. Nutritional intervention strategies for the management of overweight and obesity in primary health care: A systematic review with meta-analysis. Obes Rev. 2021 Mar;22(3):e13143. doi: 10.1111/obr.13143. Epub 2020 Oct 2. PMID 33006421
- [Background] Pereira SS, Alvarez-Leite JI. Low-Grade Inflammation, Obesity, and Diabetes. Curr Obes Rep. 2014 Dec;3(4):422-31. doi: 10.1007/s13679-014-0124-9. PMID 26626919
- [Background] Magliano D, Boyko EJ (2021) IDF diabetes atlas, 10th edition. International Diabetes Federation, Brussels
- [Background] World Obesity Day 2022 - Accelerating action to stop obesity. https://www.who.int/news/item/04-03-2022-world-obesity-day-2022-accelerating-action-to-stop-obesity. Accessed 20 Nov 2022
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646